CLINICAL TRIAL: NCT03093844
Title: Safety and Efficacy of Miltenyi CliniMACS® CD34 Reagent System for Transplant Protocol Utilizing Haploidentical CD34+ Selected Cells Combined With Single Unit Umbilical Cord Blood Transplant for Treatment of High-risk Hematologic Disorders
Brief Title: Haploidentical CD34+ Selected Cells Combined With Single Unit Umbilical Cord Blood Transplant for Treatment of High-risk Hematologic Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-1672.cc
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Hematologic Disorders
Keywords: Stem Cell Transplant; Umbilical Cord Blood Transplant; Haploidentical CD34+ Selected Cells
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Intervention Model Description: This is a phase 1/phase 2 study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Miltenyi CliniMACS® CD34 Reagent System (Experimental): The haploidentical donor will be mobilized by G-CSF and undergo one apheresis to collect CD34+ selected stem cell product after Miltenyi CliniMACS® CD34+ selection. The products will be cryopreserved until the time of transplantation.
  Recipients will receive a standard conditioning regimen. After the conditioning regimen, the subjects will receive an allograft on day 0 containing donor CD34+ cells that have been positively selected and T-cell depleted following G-CSF mobilization combined with a single UCB unit. UCB unit will not be manipulated, and will be prepared and infused separately following standard of care procedure.
  Interventions: Device: Miltenyi CliniMACS® CD34 Reagent System

INTERVENTIONS:
Device: Miltenyi CliniMACS® CD34 Reagent System — Miltenyi CliniMACS® CD34 Reagent System will be used to prepare CD34+ enriched/T-cell depleted cells from haploidentical mobilized peripheral blood.

SUMMARY:
This is a study to evaluate the safety and efficacy of Miltenyi CliniMACS® CD34 Reagent System to promote engraftment of haploidentical CD34+ selected cells combined with single unit umbilical cord blood transplant for treatment of high-risk hematologic disorders.

DETAILED DESCRIPTION:
In this clinical protocol, the CliniMACS® CD34 Reagent System will be used for processing hematopoietic progenitor cells collected by apheresis (HPC, Apheresis) from an allogeneic, HLA-haploidentical, related donor to obtain a CD34+ cell-enriched population for hematopoietic reconstitution. The haploidentical donor will be mobilized by G-CSF and undergo one apheresis to collect CD34+ stem cells. The products will be cryopreserved until the time of transplantation. Recipients with hematologic disorders who require transplant will receive a standard conditioning regimen and will receive an allograft on day 0 containing donor CD34+ cells that have been positively selected and T-cell depleted following G-CSF mobilization combined with a single UCB unit.

ELIGIBILITY:
Inclusion Criteria - Recipient

* Ages 18-80 years inclusive
* Diagnosed with high risk hematologic disorders warranting stem cell transplant per institutional standard of care
* Lack HLA-identical related donor
* Availability of at least one HLA- haploidentical (i.e. => 5/10 and <= 8/10 HLA match) related donor (HLA-A, B, C, DR, and DQ loci) who is available to donate CD34+ cells.
* Availability of at least one 4/6 HLA-matched (HLA-A, B, and DR loci) cord blood unit from the National Marrow Donor Program (NMDP). The cord blood unit must contain a minimum TNC (prior to thawing) of at least 2x107 cells per kilogram of recipient body weight
* Ability to comprehend the nature of the treatment 6.2. Exclusion Criteria - Recipient (any of the following)
* HLA identical (6/6) related donor available and readily accessible at time of transplantation evaluation
* Any patient not meeting institutional standard guidelines for transplant eligibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2025-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Gutman, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Besien K, Childs R. Haploidentical cord transplantation-The best of both worlds. Semin Hematol. 2016 Oct;53(4):257-266. doi: 10.1053/j.seminhematol.2016.07.004. Epub 2016 Jul 25. PMID 27788764
- [Background] van Besien K, Koshy N, Gergis U, Mayer S, Cushing M, Rennert H, Reich-Slotky R, Mark T, Pearse R, Rossi A, Phillips A, Vasovic L, Ferrante R, Hsu YM, Shore T. Cord blood chimerism and relapse after haplo-cord transplantation. Leuk Lymphoma. 2017 Feb;58(2):288-297. doi: 10.1080/10428194.2016.1190970. Epub 2016 Jun 23. PMID 27333804
- [Background] Magro E, Regidor C, Cabrera R, Sanjuan I, Fores R, Garcia-Marco JA, Ruiz E, Gil S, Bautista G, Millan I, Madrigal A, Fernandez MN. Early hematopoietic recovery after single unit unrelated cord blood transplantation in adults supported by co-infusion of mobilized stem cells from a third party donor. Haematologica. 2006 May;91(5):640-8. PMID 16670070
- [Background] Kwon M, Bautista G, Balsalobre P, Sanchez-Ortega I, Serrano D, Anguita J, Buno I, Fores R, Regidor C, Garcia Marco JA, Vilches C, de Pablo R, Fernandez MN, Gayoso J, Duarte R, Diez-Martin JL, Cabrera R. Haplo-cord transplantation using CD34+ cells from a third-party donor to speed engraftment in high-risk patients with hematologic disorders. Biol Blood Marrow Transplant. 2014 Dec;20(12):2015-22. doi: 10.1016/j.bbmt.2014.08.024. Epub 2014 Sep 22. PMID 25255162

RESULTS

PARTICIPANT FLOW:
Groups:
- Miltenyi CliniMACS® CD34 Reagent System: The haploidentical donor will be mobilized by G-CSF and undergo one apheresis to collect CD34+ selected stem cell product after Miltenyi CliniMACS® CD34+ selection. The products will be cryopreserved until the time of transplantation.
  Recipients will receive a standard conditioning regimen. After the conditioning regimen, the subjects will receive an allograft on day 0 containing donor CD34+ cells that have been positively selected and T-cell depleted following G-CSF mobilization combined with a single UCB unit. UCB unit will not be manipulated, and will be prepared and infused separately following standard of care procedure.
  Miltenyi CliniMACS® CD34 Reagent System: Miltenyi CliniMACS® CD34 Reagent System will be used to prepare CD34+ enriched/T-cell depleted cells from haploidentical mobilized peripheral blood.
Period: Overall Study
Arm/Group | Miltenyi CliniMACS® CD34 Reagent System
Started | 150
Completed | 150
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 150 participants treated. 146 alive at D42 to analyze primary outcome results.
Arm/Group | Miltenyi CliniMACS® CD34 Reagent System
Number analyzed (Participants) | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 125
  >=65 years | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 126
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With Successful Engraftment
Description: To determine the rate of successful engraftment of patients who received haploidentical CD34+ selected cells combined with single unit umbilical cord blood transplant. Failure defined as failure of Miltenyi CliniMACS® CD34 Reagent System to select CD34+ cells, and/or failure to engraft by day 42.
Time Frame: 42 days
Population: Participants who were eligible, received cell product, and were alive at D42.
Measure: Count of Participants; unit: Participants
Arm/Group | Miltenyi CliniMACS® CD34 Reagent System
Number analyzed (Participants) | 146
Participants | 144

ADVERSE EVENTS:
Time Frame: Until engraftment (approximately 42 days).
Arm/Group | Miltenyi CliniMACS® CD34 Reagent System
All-Cause Mortality (participants affected / at risk) | 4/150
Serious Adverse Events (participants affected / at risk) | 2/150
Other Adverse Events (participants affected / at risk) | 0/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Miltenyi CliniMACS® CD34 Reagent System (N=150)
General disorders and administration site conditions - Other, specify (General disorders) | 2 (2) — Failure to engraft by day 42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT03093844/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT03093844/ICF_001.pdf